CLINICAL TRIAL: NCT05478044
Title: Effect of Ascorbic Acid as a Final Flush on Post-operative Pain After Single Visit Root Canal Treatment for Patients With Symptomatic Irreversible Pulpits Related to Mandibular Molars: Randomized Controlled Trial.
Brief Title: Effect of Ascorbic Acid Final Flush on Post-operative Pain in Mandibular Molars.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Kariman Mohammed Mohammed Amin Ismaiel, Research assistant of endodontics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ENDO 3 - 7 - 1
Record Dates: First submitted 2022-07-24; First posted 2022-07-28 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Ascorbic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ascorbic acid (Experimental): Ascorbic acid IV ampoules 20% as a final flush irrigation 3ml after cleaning and shaping.
  Interventions: Drug: Ascorbic acid
- Saline (Placebo Comparator): A mixture of sodium chloride and water (0.9%) as a final flush irrigation 3 ml after cleaning and shaping.
  Interventions: Other: saline

INTERVENTIONS:
Drug: Ascorbic acid — Ascorbic acid IV ampoules (20%).
  Other Names: Vitamin C
  Arms: Ascorbic acid
Other: saline — saline (0.9%)
  Arms: Saline

SUMMARY:
The study is conducted to evaluate the effect of Ascorbic acid as a final flush on post operative pain after single visit root canal treatment in cases with symptomatic irreversible pulpits.

ELIGIBILITY:
Inclusion Criteria:

* Patients above 18 years old and to 60.
* Male or female.
* Patients seeking root canal treatment.
* mandibular molar teeth with symptomatic irreversible pulpits with preoperative acute or moderate pain with hot and cold stimulation with normal periapical radiographic appearance .
* healthy patient (ASA I,II).
* Patient who can understand NRS and sign informed consent.

Exclusion Criteria:

* Medically compromised patients having significant systemic disorders. (ASA III or IV).
* History of intolerance to NSAIDS.
* External root resorption.
* Internal root resorption.
* Vertical root fracture.
* Periapical lesion.
* Pregnancy.
* Use of ibuprofen in the last 12 hour.
* Bleeding disorder.
* Long term corticosteroid use.
* Mobility Grade II or III.
* Pocket depth more than 5mm.
* Previous root canal therapy.
* Non-restorability.
* TMJ problems, bruxism, clenching or traumatic occlusion.
* Inability to perceive the given instructions.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Pain intensity measured by numerical rating scale where 0= no pain, 1-3= mild pain, 4-6= moderate pain and 7-10= severe pain. | up to 48 hours after root canal treatment.

SECONDARY OUTCOMES:
If there are analgesics taken by the patient after root canal treatment and that will be measured by a questionnaire. | up to 48 hours.